CLINICAL TRIAL: NCT02258204
Title: Effets de la kétamine en Association Avec le Rt-PA au Cours de l'Infarctus cérébral Aigu: étude Pilote contrôlée randomisée en Double Aveugle Avec critère de Jugement Radiologique
Brief Title: Ketamine for Thrombolysis in Acute Ischemic Stroke
Acronym: KETA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Société Française d'Anesthésie Réanimation (Unknown); Fondation NRJ (Unknown)
Responsible Party: Principal Investigator, Emmanuel TOUZE, Professor, University Hospital, Caen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KETA
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Stroke
Keywords: Cerebral Infarct; Thrombolysis; Tissue-type plasminogen activator; Neuroprotection; Anesthetic agent; Magnetic resonance imaging
MeSH Terms: conditions — Stroke; Cerebral Infarction | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tPA-placebo (Placebo Comparator): tPA infusion : 0.9 mg/kg (90 mg maximum), 10% of the total dose is administered as an initial IV bolus dose over 1 minute and the remainder of the dose is infused over 60 minutes.
  Saline infusion : 0.15 mL/kg IV bolus (maximum 15 mL) followed by an IV infusion of 0.15 mL/kg over 60 minutes (maximum 15 mL).
  Interventions: Drug: Placebo
- tPA-ketamine (Experimental): tPA infusion : 0.9 mg/kg (90 mg maximum), 10% of the total dose is administered as an initial IV bolus dose over 1 minute and the remainder of the dose is infused over 60 minutes.
  Ketamine infusion : 0.15 mg/kg IV bolus (maximum 15 mg) followed by an IV infusion of 0.15 mg/kg over 60 minutes (maximum 15 mg).
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Co-administration of subanesthetic dose of ketamine with tPA for thrombolysis in acute ischemic stroke.
  Arms: tPA-ketamine
Drug: Placebo
  Arms: tPA-placebo

SUMMARY:
KETA trial is a nonprofit, double-blind, randomized, controlled pilot trial with aiming to determine if co-administration of ketamine with recombinant of tissue type plasminogen activator (tPA) for thrombolysis in acute ischemic stroke compared with tPA co-administered with placebo, decreases cerebral infarction growth in diffusion weighted imaging between admission and day 1. Eligibility applies to patients with symptomatic ischemic stroke seen within 4.5 h of onset with middle cerebral artery or distal internal carotid artery occlusion, no contraindication to intravenous tPA-mediated thrombolysis and eligible to endovascular treatment of stroke (i.e. thrombectomy). The study has been designed to have 80% power to detect a 80% decrease of infarct volume growth in the tPA-ketamine group at a two-sided type I error rate of 5%. For this purpose, at least 25 patients per arm should be enrolled.

DETAILED DESCRIPTION:
Rationale - Tissue-type plasminogen activator (tPA) is a double-sided molecule, with beneficial effect in acute ischemic stroke due to its intravascular fibrinolytic activity but with potential deleterious effect due to its ability to potentiate neuronal N-methyl-D-aspartate (NMDA) receptor signalling (Nicole et al., 2001). Co-administration of sub-anesthetic dose of ketamine - a non-competitive inhibitor of NMDA receptor - was shown to improve efficacy of tPA-mediated thrombolysis following stroke in rodents (Gakuba et al, 2011).

Aims - To assess efficacy and safety of co-administration of ketamine with tPA compared with tPA-placebo infusion in patients with acute ischemic stroke.

Sample size estimates -With 25 patients per group, the trial has a 80% probability of detecting a 80% decrease of infarct volume growth in the tPA-ketamine group compared with the tPA-placebo group on day 1 after admission at a two-sided type I error rate of 5%.

Study outcomes - The primary efficacy outcome is cerebral infarction growth on diffusion weighted imaging between admission and day 1. The primary safety measure is mortality and/or symptomatic intracerebral hemorrhage rate at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Sudden focal neurological deficit attributable to acute ischemic stroke.
* Age between 18 and 85.
* Time from symptom onset less than 4.5 hours.
* NIHSS score between 7 and 20.
* Informed consent for participation.
* Ketamine can be administered within 15 minutes after onset of tPA infusion.
* MRI-based AIS diagnosis.
* Middle cerebral (M1 or M2 segment) and/or distal internal carotid artery occlusion.
* No intracranial hemorrhage on MRI.
* Patient eligible for thrombectomy.

Exclusion Criteria:

* Contraindication to IV tPA treatment.
* Contraindication to ketamine.
* Contraindication to MRI.
* Contraindication to intravascular iodinated contrast media.
* Consciousness level >1 on question 1a of NIHSS.
* Pre-stroke mRS ≥3.
* Concomitant medical illness that would interfere with outcome assessments and follow-up (e.g. advanced cancer or respiratory disease).
* Previous participation in this trial or current participation in another investigational drug trial.
* Infarct volume on diffusion weighted MRI more than 100 mL.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cerebral infarction growth on diffusion weighted magnetic resonance imaging between admission and day 1. | Day 1

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale | day 0, day 1, day 7 and day 90
Modified Rankin Scale | day 90
Infarction volume on diffusion weighted magnetic resonance imaging | day 1
T2-weighted Fluid Attenuated Inversion Recovery Imaging infarct volume | day 90
Symptomatic intracerebral hemorrhage and/or death | day 90
Arterial patency | day 0 (before and after thrombectomy) and day 1
  Arterial patency will be assessed with the Thrombolysis in Cerebral Infarction (TICI) Score on day 0 before and after thrombectomy (digital subtraction angiography) and day 1 (magnetic resonance angiography).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen, Caen, France

REFERENCES:
- [Background] Nicole O, Docagne F, Ali C, Margaill I, Carmeliet P, MacKenzie ET, Vivien D, Buisson A. The proteolytic activity of tissue-plasminogen activator enhances NMDA receptor-mediated signaling. Nat Med. 2001 Jan;7(1):59-64. doi: 10.1038/83358. PMID 11135617
- [Background] Gakuba C, Gauberti M, Mazighi M, Defer G, Hanouz JL, Vivien D. Preclinical evidence toward the use of ketamine for recombinant tissue-type plasminogen activator-mediated thrombolysis under anesthesia or sedation. Stroke. 2011 Oct;42(10):2947-9. doi: 10.1161/STROKEAHA.111.620468. Epub 2011 Aug 4. PMID 21817137